CLINICAL TRIAL: NCT02927288
Title: Identifying Biomarkers That Distinguish Post-Traumatic Stress Disorder and Mild Traumatic Brain Injury Using Advanced Magnetic Resonance Spectroscopy
Brief Title: Identifying Biomarkers That Distinguish PTSD and mTBI Using Advanced Magnetic Resonance Spectroscopy
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lin, Alexander P.,Ph.D., Director of the Center for Clinical Spectroscopy, Brigham and Women's Hospital
Other Study IDs: W81XWH-10-1-0785
Record Dates: First submitted 2016-09-30; First posted 2016-10-07 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Post-Traumatic Stress Disorders; Brain Injuries
Keywords: PTSD, mTBI
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Military subjects with mTBI: mTBI/concussion only Group: Participants must have been clinically diagnosed with mTBI/concussion according to criteria outline by the World Health Organization (WHO; Holm et al., 2005) and be at least three month post-injury. Participants in the mTBI/concussion only group must not have a concurrent diagnosis of PTSD and must score below 25 on the Post-traumatic stress Check List for Civilians (PCL-C).
- Military subjects with PTSD: Participants in the PTSD only group must have a clinical diagnosis of PTSD, following criteria outlined in the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV TR). Proof of diagnosis will be obtained from participants via a request for release of pertinent medical records. Participants in this group must not have a history of mTBI or concussion.
- Military subjects with mTBI and PTSD: Participants in the mixed group must meet criteria for mTBI/concussion and PTSD as outlined above.
- Military healthy control: Participants in the military control group will meet all general requirements for participation but will not have a history of either mTBI/concussion or PTSD, as described above. Participants in this group will include service members on Active Duty and those currently serving with National Guard or Reserve forces.
- Civilian healthy control: Participants in the civilian control group will meet all general requirements for participation but will not have a history of either mTBI/concussion or PTSD, as described above.

SUMMARY:
The purpose of this study is to develop a new test to help diagnose mild traumatic brain injury (mTBI) and post-traumatic stress disorder (PTSD) in soldiers. Chemicals in the brain will be measured using a Magnetic Resonance Spectroscopy (MRS) scan. In the study, the investigators will compare the information they obtain from scans of participants with mTBI, PTSD or both, to scans from healthy volunteers to understand the differences between these groups. If the results can tell the difference between participants with mTBI and PTSD, the investigators should be able to help safely diagnose patients in the future.

DETAILED DESCRIPTION:
Soldiers from the US Army, with well characterized diagnosis of mTBI or PTSD, will be recruited in the first year as will age-matched healthy controls from the military and civilian populations. MRI, single voxel MRS, and two-dimensional correlated spectroscopy (2D COSY) MRS will be acquired from each participant at the Brigham and Women's Hospital (BWH). This data will be anonymized and transferred to the Draper Laboratories. Biomarkers for each disease will be identified by comparison with control data. These biomarkers will then be fed into classifiers that will then be validated with a similar cohort acquired in the second year. The second cohort of subjects will then be incorporated into the classifier algorithms for a stronger and more robust classification from which a diagnostic test will emerge. To test this diagnostic evaluation the data analysis by both BWH and Draper labs will be blinded to the characterization of the participants and from the MRS results, the investigators will predict if the participant has mTBI, PTSD, both, or neither. Finally, all data will then be fused into the algorithms to provide a final classifier. The results of the final classifier will then be correlated with clinical, neuropsychological, and neuroanatomical indices of mTBI and PTSD. These correlations will provide the most complete biochemical analysis of mTBI and PTSD which may lead to insight into alternate pathways for drug development.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 55
2. Male and female
3. High School diploma or General Educational Development (GED) equivalent

Exclusion Criteria:

1. History of brain tumor, epilepsy, dementia, and other neurological disorders
2. History of psychotic, bipolar, or other mental disorder aside from PTSD
3. Substance abuse and/or use within the past month of skeletal muscle relaxants, narcotics, anticonvulsants, neuroleptics, benzodiazepines, cerebral stimulants, sedatives, or hypnotics during the month prior to testing, or a "dirty" urine specimen (i.e., containing amphetamines, barbiturates, cocaine, opiates, benzodiazepines, methaqualone, propoxyphene, phencyclidine, methadone, or cannabinoids)
4. Alcohol use 24 hours prior to testing. Subjects will be asked to abstain 24 hours in advance as alcohol can be detected in the MRS spectrum as a multiplet at 1.5 ppm.
5. Inability to give informed consent for participation
6. Any contraindications for MR imaging and spectroscopy

   1. electrical implants such as cardiac pacemakers or perfusion pumps
   2. ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants
   3. ferromagnetic objects such as jewelry or metal clips in clothing
   4. any greater than normal potential for cardiac arrest
   5. pregnancy (female of childbearing age and are still having your menstrual periods will be asked to give a urine sample for a pregnancy test that will be administered by the technologist).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 330 men and women from the Massachusetts National Guard, Active Duty Army, and veterans in the New England area and Brigham and Women's Hospital, Boston as well as healthy military and civilians will take part in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
NAA to Creatine (NAA/Cr) Ratio (no units) | One year
  NAA/Cr ratio is a neuronal marker. The average of NAA/Cr ratios for all five groups are the following:
  civilian control 1.37 military control 1.38 military TBI 1.33 military PTSD 1.34 military mTBI and PTSD 1.42

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Lin, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Data may be uploaded to FITBIR in the future.